CLINICAL TRIAL: NCT04944771
Title: An Open-label, Randomized, Crossover Study in Healthy Subjects to Evaluate the Effect of Food and Acid Reducing Agent(s) on the Pharmacokinetics of Capivasertib
Brief Title: Study to Assess the Effect of Food and Acid Reducing Agents on the Absorption of Capivasertib in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D3614C00005; 2021-000836-74 (EudraCT Number)
Record Dates: First submitted 2021-06-28; First posted 2021-06-30 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Solid and Hematological Malignancies
Keywords: Crossover; Acid reducing agent; Food effect; Pharmacokinetics; Serine/threonine specific protein kinase inhibitor
MeSH Terms: conditions — Hematologic Neoplasms | interventions — capivasertib; Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Treatment ABC (Experimental): Participants will be randomized to receive oral doses of Treatment A, Treatment B and Treatment C.
  Interventions: Drug: Capivasertib; Drug: Rabeprazole
- Treatment ACB (Experimental): Participants will be randomized to receive oral doses of Treatment A, Treatment C and Treatment B.
  Interventions: Drug: Capivasertib; Drug: Rabeprazole
- Treatment BAC (Experimental): Participants will be randomized to receive oral doses of Treatment B, Treatment A and Treatment C.
  Interventions: Drug: Capivasertib; Drug: Rabeprazole
- Treatment BCA (Experimental): Participants will be randomized to receive oral doses of Treatment B, Treatment C and Treatment A.
  Interventions: Drug: Capivasertib; Drug: Rabeprazole
- Treatment CAB (Experimental): Participants will be randomized to receive oral doses of Treatment C, Treatment A and Treatment B.
  Interventions: Drug: Capivasertib; Drug: Rabeprazole
- Treatment CBA (Experimental): Participants will be randomized to receive oral doses of Treatment C, Treatment B and Treatment A.
  Interventions: Drug: Capivasertib; Drug: Rabeprazole
- Treatment DEF (Experimental): Participants will be randomized to receive oral doses of Treatment D, Treatment E and Treatment F.
  Interventions: Drug: Capivasertib
- Treatment DFE (Experimental): Participants will be randomized to receive oral doses of Treatment D, Treatment F and Treatment E.
  Interventions: Drug: Capivasertib
- Treatment EDF (Experimental): Participants will be randomized to receive oral doses of Treatment E, Treatment D and Treatment F.
  Interventions: Drug: Capivasertib
- Treatment EFD (Experimental): Participants will be randomized to receive oral doses of Treatment E, Treatment F and Treatment D.
  Interventions: Drug: Capivasertib
- Treatment FDE (Experimental): Participants will be randomized to receive oral doses of Treatment F, Treatment D and Treatment E.
  Interventions: Drug: Capivasertib
- Treatment FED (Experimental): Participants will be randomized to receive oral doses of Treatment F, Treatment E and Treatment D.
  Interventions: Drug: Capivasertib

INTERVENTIONS:
Drug: Capivasertib — Participants will receive single oral dose of capivasertib on Day 1 for Treatments A, B, C, D, E and F.
Drug: Rabeprazole — Participants will receive twice daily oral doses of rabeprazole for 3 days (Days -3 to -1) and a single dose on the morning of Day 1 for Treatment C.
  Arms: Treatment ABC; Treatment ACB; Treatment BAC; Treatment BCA; Treatment CAB; Treatment CBA

SUMMARY:
This is a two-part, open-label, randomized, crossover study in healthy subjects (vasectomized males and women of non-childbearing potential), performed at 2 study centers

DETAILED DESCRIPTION:
Part 1 of the study will comprise:

* A screening period of maximum 28 days.
* Three treatment periods [Treatment A: Single oral dose of capivasertib in overnight fasted state, Treatment B:Single oral dose of capivasertib in fed state (high-fat, high-calorie breakfast) and Treatment C:Twice daily oral doses of rabeprazole for 3 days and a single dose on Day 1, and a single oral dose of capivasertib in fasted conditions] during which subjects will be resident from the morning of Day -1 (Day -4 for subjects receiving rabeprazole [Treatment C]) and discharged after the last pharmacokinetic (PK) sample collection, 48 hours after dosing of capivasertib of each treatment period.
* A final visit 7 to 14 days after the last capivasertib PK sample in Treatment Period 3.

Part 2 of the study will only be initiated if the findings from Part 1 show an interaction or are inconclusive. Part 2 of the study will comprise:

* A screening period of at least 28 days.
* Three treatment periods [Any 3 treatments: Treatment D:Single oral dose of capivasertib in overnight fasted state, Treatment E: Single oral dose of capivasertib in fed state (low-fat, low-calorie breakfast), Treatment F: Single oral dose of capivasertib in partially fasted conditions (food restricted from 2 hours prior to dosing until 1 hour after dosing), Treatment G: Single oral dose of capivasertib and single dose of famotidine in fasted condition and Treatment H: Twice daily oral doses of rabeprazole for 3 days (Days -3 to -1) and a single oral dose of capivasertib in fed state] during which subjects will be resident from the morning of Day -1 (Day -4 for subjects receiving rabeprazole [Treatment H]) and will be discharged after the last PK sample collection 48 hours after dosing of capivasertib of each treatment period.
* A final visit 7 to 14 days after the last capivasertib PK sample in Treatment Period 3.

The interim results from Part 1 indicated a potentially clinically relevant food interaction only and therefore Treatments D, E, and F will be studied in Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Healthy male and female subjects aged 18 to 58 years with suitable veins for cannulation or repeated venipuncture.
* Females must not be lactating and must be of non-childbearing potential, confirmed at screening:

  1. Postmenopausal defined as aged > 40 years and amenorrhea for at least 12 months or more following cessation of all exogenous hormonal treatments and follicle stimulating hormone levels in the postmenopausal range.
  2. Documentation of irreversible/permanent surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation, at least 6 months prior to screening.
* Male subjects must be vasectomized, at least 6 months prior to screening, with documented post-procedural medical assessment of surgical success.
* Have a body mass index between 18.0 and 29.9 kg/m^2 (inclusive) for males and 18 to 32 kg/m^2 (inclusive) for females; and weigh at least 50 kg and no more than 100 kg inclusive.
* Non-smoker, defined as a subject who has not smoked previously or who has discontinued smoking.

Exclusion Criteria:

* History of any clinically significant disease or disorder.
* History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of investigational medicinal product (IMP).
* Any clinically significant abnormal findings in vital signs at screening and/or admission to the study center.
* Clinically significant abnormalities in glucose metabolism defined by any of the following:

  1. Diagnosis of diabetes mellitus type I or II (irrespective of management).
  2. Blood glucose value ≥ 5.9 mmol/L after fasting for at least 8 hours, at screening or on admission to study center.
  3. Glycosylated hemoglobin > upper limit of normal (up to 6.2% [44 mmol/mol]).
* Any positive result on screening for serum hepatitis B surface antigen or antibody to hepatitis B core antigen, hepatitis C antibody, and human immunodeficiency virus antibody.
* Known or suspected history of drug abuse.
* Has received another new chemical entity within 3 months of the first administration of IMP in this study.
* Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to screening.
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator or history of hypersensitivity to drugs with a similar chemical structure or class to capivasertib, rabeprazole, or famotidine.
* Subjects who have previously received capivasertib.
* Subject has a positive test result for Severe acute respiratory syndrome coronavirus 2 reverse transcription polymerase chain reaction on admission.
* Subject has clinical signs and symptoms consistent with Coronavirus Disease 2019 (COVID-19) (eg, fever, dry cough, dyspnea, sore throat, anosmia/hyposmia, loss or reduced taste, and fatigue) or confirmed infection by appropriate laboratory test within the last 4 weeks prior to screening or on admission.
* History of severe COVID-19 (hospitalization, extracorporeal membrane oxygenation, mechanically ventilated).
* Subjects who are regularly exposed to the risk of COVID-19 infection as part of their daily life (eg, health care professionals working in COVID-19 wards or at emergency departments).
* Subjects who have had a COVID-19 vaccine within 3 weeks prior to screening or are planning to get a COVID-19 vaccine during the study.

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-04 (Actual)

PRIMARY OUTCOMES:
Cmax of Capivasertib | Part 1 and Part 2: From Day 1 to Day 3
  Maximum observed plasma (peak) drug concentration (Cmax) of capivasertib when administered alone under fed and fasted conditions, and in combination with acid reducing agent(s) rabeprazole and famotidine (if required).
AUCinf of Capivasertib | Part 1 and Part 2: From Day 1 to Day 3
  Area under plasma concentration time curve from zero to infinity (AUCinf) of capivasertib when administered alone under fed and fasted conditions, and in combination with acid reducing agent(s) rabeprazole and famotidine (if required).
AUClast of Capivasertib | Part 1 and Part 2: From Day 1 to Day 3
  Area under the plasma concentration curve from zero to the last quantifiable concentration (AUClast) of capivasertib when administered alone under fed and fasted conditions, and in combination with acid reducing agent(s) rabeprazole and famotidine (if required).

SECONDARY OUTCOMES:
Number of participants with serious and non-serious adverse events | Part 1: From Screening (Day -28 to Day -5) upto Follow-up Visit/Early Termination (7 to 14 days); Part 2: From Screening (Day -28 to Day -2) upto Follow-up Visit/Early Termination (7 to 14 days)
  Safety and tolerability of capivasertib when administered alone under fed and fasted conditions, and in combination with acid reducing agent(s) rabeprazole and famotidine (if required).

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home